CLINICAL TRIAL: NCT03264937
Title: Randomized Evaluation of Social-software Improving Warfarin Therapy in Patients With Mechanical Heart Valve Replacement
Brief Title: Social-software iMproving wARfarin Therapy
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Litao Zhang, MD, Manager of anticoagulation clinic, Wuhan Asia Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-P-033
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Anticoagulants Causing Adverse Effects in Therapeutic Use; Patient Compliance
Keywords: TTR; INR; Warfarin; social software
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social-software management group (Experimental): We set up a mini-program based on wechat application. We instruct warfarin therapy via social-software including dose adjustment, answer questions, remind monitoring INR et.al.
  Interventions: Behavioral: Social-software management
- Routine management group (No Intervention): This is the control group, Warfarin therapy was managed via traditional style without social software intervention.

INTERVENTIONS:
Behavioral: Social-software management — Using Wechat application, a social platform, to manage warfarin therapy in patients with mechanical valve replacement.
  Arms: Social-software management group

SUMMARY:
Poor anticoagulation quality is a major problem among Chinese patients receiving warfarin therapy in traditional health care settings. Improving warfarin therapy has been crucial for Chinese patients. Wechat is social-software in China. Most of all Chinese adults use Wechat, as well as our patients. So we set up a Wechat-based mini-program to instruct Chinese patients' warfarin therapy. We aim to assess whether social software could improve warfarin therapy in Chinese patients by conducting a single-centre, open-label, prospective, randomized clinical trial.

DETAILED DESCRIPTION:
Social software is becoming a necessary of life. Wechat, powered by Tencent company, is the most popular social software in China. People can chat with others no matter how far away from each other.

Anticoagulation Quality is very important for patients receiving warfarin anticoagulation therapy, which is usually evaluated Time in therapeutic range (TTR). It is reported that TTR is very low (38.8%) in China patients. So we are planning to introduce the social software to set up a bridge for clinicians and their patients, to instruct warfarin therapy. We aim to investigate whether social software could be used to improve warfarin anticoagulation quality of Chinese patients.

We planned to enrol enough eligible patients receiving warfarin therapy due to the mechanical valves in a randomized controlled trial. Warfarin-treated patients were assigned to social software management group ( in which warfarin therapy was guided via the social platform by experienced clinicians) or to the traditional management control group (in which warfarin therapy was managed with traditional model). The primary outcomes the first time to bleeding or thrombotic events, the secondary outcomes were an elevation in time in therapeutic range (TTR) of international normalized ratio (INR), reduction in INR variation and number of extremely high INR results during 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Received mechanical valve replacement;
* Receiving warfarin anticoagulation therapy;
* Have smartphone and Know how to use wechat application and our mini-program;
* be expected to survive for the duration of the study;
* not be suffering from intracranial bleeding (intracranial haemorrhage, subarachnoid haemorrhage, hemorrhagic stroke) or any other contraindication described in the warfarin package insert;
* be willing to be randomized;
* sign the informed consent form;
* not be enrolled in another randomized clinical trial that involves a drug or device intervention.

Exclusion Criteria:

* subject has had an intracranial haemorrhage, subarachnoid haemorrhage, hemorrhagic stroke, or any other absolute/major contraindication described in the warfarin package insert within the last month
* subject enrolled in another randomized clinical trial that involves a drug or device intervention
* subject is not able to follow the protocol and all related instructions and does not have a caregiver with these skills
* Patients were considered being not suitable for this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Time to First Event | Up to 18 months
  Thrombotic events, such as Valve thrombosis, Stroke, Peripheral embolism; Major bleeding, such as cerebral hemorrhage，gastrointestinal bleeding etc.

SECONDARY OUTCOMES:
Time in therapeutic range | Up to 18 months
  Time in target range (TTR) based on Prothrombin Time standardized to the International Normalized Ratio
Individual variation of International Normalized Ratio (INR) | Up to 18 months
  Standard deviation (SD) of individual INR results
Times of extremely high International Normalized Ratio (INR) values | Up to 18 months
  Times of INR results above 4.0; Times of INR results above 12.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlu Zhang, MD,PhD, Study Director — Wuhan Asia Heart Hospital
Locations (1):
- WAHH, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
We are going to make individual participant data (IPD) available to other researchers after our paper published
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Zhang L, Li S, Li Z, Yu D, Wu H, Hua B, Xie L, Yuan X, Li Y, Zhang Z, Long Y. Social App to Improve Warfarin Therapy in Post-MHVR Chinese Patients: A Randomized Controlled Trial. Cardiovasc Ther. 2023 Jan 14;2023:2342111. doi: 10.1155/2023/2342111. eCollection 2023. PMID 36714197